CLINICAL TRIAL: NCT03092973
Title: Carotid Intima Media Thickness in Patients With Epistaxis: a Surrogate Marker for Generalised Atherosclerosis
Brief Title: Carotid Intima Media Thickness (CIMT) in Epistaxis
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: CIMT in Epistaxis
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Epistaxis; Atherosclerosis
MeSH Terms: conditions — Epistaxis; Atherosclerosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epistaxis Group
  Interventions: Diagnostic Test: Ultrasound
- Control Group
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound

SUMMARY:
Epistaxis is a very frequent emergency among adults and often needs specialised treatment in an ENT-department. Among others, atherosclerosis is often named as a reason for an increased risk for Epistaxis. To evaluate whether or not this is the case, the investigators examined the carotid intima media thickness via ultrasound in patients who were treated in the ENT-department of the University Hospital of Zurich.

ELIGIBILITY:
Inclusion Criteria:

* active or very recently active anterior or posterior epistaxis
* at least 18 years old

Exclusion Criteria:

* posttraumatic or postoperative epistaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with epistaxis and 50 healthy controls.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Carotid Intima Media Thickness in Epistaxis vs. Controls | June 2017

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soyka, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
The participant data will no longer be used by us or other researchers after the project is finished.

REFERENCES:
- [Derived] Kunz SM, Holzmann D, Soyka MB. Association of epistaxis with atherosclerotic cardiovascular disease. Laryngoscope. 2019 Apr;129(4):783-787. doi: 10.1002/lary.27604. Epub 2018 Dec 13. PMID 30549051